CLINICAL TRIAL: NCT03919942
Title: Effect of Oxyflower® Gel as a Coadjuvant in Pericoronitis Treatment: Controlled Randomized Clinical Trial
Brief Title: Effect of Oxyflower® Gel as a Coadjuvant in Pericoronitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16042019
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Pericoronitis
Keywords: Quality of life; Pericoronitis; Phytotherapy
MeSH Terms: conditions — Pericoronitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OxyFlower gel (Experimental): pericoronitis treatment with oxyflower gel.
  Interventions: Other: OxyFlower gel
- Chlorhexidine gel (Experimental): pericoronitis treatment with chlorhexidine gel.
  Interventions: Other: Chlorhexidine gel
- Placebo gel (Placebo Comparator): pericoronitis treatment with placebo gel.
  Interventions: Other: Placebo gel

INTERVENTIONS:
Other: OxyFlower gel — the region with pericoronitis was debrided using gauze and curettes, with copious irrigation with sterile saline solution. At this moment, the gel was applied topically under the pericoronal hood, with a standard volume of 2microIiters, using a dosing syringe. Then, participants received instructions on oral hygiene and how to use the gel at home, twice a day for one week. After 30 days, it was performed third molar removal or distal wedge removal
  Arms: OxyFlower gel
Other: Chlorhexidine gel — the region with pericoronitis was debrided using gauze and curettes, with copious irrigation with sterile saline solution. At this moment, the gel was applied topically under the pericoronal hood, with a standard volume of 2microIiters, using a dosing syringe. Then, participants received instructions on oral hygiene and how to use the gel at home, twice a day for one week. After 30 days, it was performed third molar removal or distal wedge removal.
  Arms: Chlorhexidine gel
Other: Placebo gel — the region with pericoronitis was debrided using gauze and curettes, with copious irrigation with sterile saline solution. At this moment, the gel was applied topically under the pericoronal hood, with a standard volume of 2microIiters, using a dosing syringe. Then, participants received instructions on oral hygiene and how to use the gel at home, twice a day for one week. After 30 days, it was performed third molar removal or distal wedge removal
  Arms: Placebo gel

SUMMARY:
The objective of this study is to evaluate the clinical effect and the impact on the quality of life of the coadjuvant treatment with Oxyflower® gel in cases of pericoronitis in lower third molar, compared to chlorhexidine gel and placebo gel.

DETAILED DESCRIPTION:
This study consist of 51 participants diagnosed with pericoronitis who received coadjuvant treatment with gel. The participants were submitted to emergency treatment, with local debridement and irrigation with saline solution followed by topical application of the randomized gel: oxyflower®, chlorhexidine, or placebo gel. In cases of pericoronitis with systemic signs / symptoms, such as fever, malaise and lymphadenopathy, systemic antibiotic therapy was prescribed one hour before debridement, lasting seven days. All participants received oral hygiene guidelines and were instructed to apply the same gel twice daily for one week . After 30 days, it was performed tooth removal for cases in which there is not enough space for dental eruption; or distal wedge surgery when there is space for dental eruption with excessive gingiva in the distal. It was evaluated as outcomes: pain, quality of life, depth of probing, level of bone crest in the distal of second molar, buccal opening and extent of edema / erythema. A comparative analysis was performed between the groups, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* signs / symptoms of pericoronitis with
* spontaneous pain
* ASA I or II
* Consent to participate

Exclusion Criteria:

* Periodontal status level IV
* Smokers
* antibiotic therapy in the last 2 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quality of life | baseline, 30 days
  Oral health related quality of life measured by questions related to the quality of life. This questionnaire comprises 14 items within 7 subscales (functional limitation, pain, psychological discomfort, physical disability, psychological disability, social disability, deficit).
Change from Baseline Pain | baseline, 1,3,7,15 and 30 days
  Post-operative pain measured by visual analogic scale (VAS). The VAS comprises a 10cm horizontal line, with no marks. When responding to a VAS, subjects specify their level of pain by indicating a position along a continuous line between two end-points. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Change from Baseline trismus | baseline, 1,3,7,15 and 30 days
  maximum mouth opening measured as maximum distance between incisal edges of upper and lower central incisors.
change from edema / erythema | baseline, 1, 3, 7, 15 and 30 days
  The extent of edema / erythema was assessed by measuring the greater vestibulo-lingual and mesio-distal distance of the lesion, by periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia F Gonçalves, PhD, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No